CLINICAL TRIAL: NCT03294330
Title: SPY-X: A Study to Assess the Feasibility of Using Real-time Fluorescence Lymphangiography Alone for Sentinel Node Localization in Patients With Melanoma or Breast Cancer
Brief Title: SPY-X: A Study to Assess the Feasibility of Using SPY Alone for Sentinel Node Localization for Melanoma or Breast Cancer
Acronym: SPYX
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Milton S. Hershey Medical Center (Other)
Collaborators: Vassar Brothers Medical Center (Other); Emory University (Other)
Responsible Party: Principal Investigator, Colette Pameijer, Medical Doctor, Milton S. Hershey Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 7046
Record Dates: First submitted 2017-09-22; First posted 2017-09-27 (Actual); Results first posted 2023-01-12 (Actual); Last update posted 2023-01-12 (Actual); Status verified 2022-12

CONDITIONS: Sentinel Lymph Node; Melanoma (Skin); Breast Cancer
MeSH Terms: conditions — Melanoma; Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Patients with Melanoma or Breast Cancer (Experimental): The SPY machine used in conjunction with the IC-green kit will be used exclusively to identify sentinel nodes in patients diagnosed with Melanoma or Breast Cancer who are undergoing sentinel lymph node biopsy.
  Interventions: Drug: IC-Green KIT

INTERVENTIONS:
Drug: IC-Green KIT — fluorescence lymphangiography with the use of IC-Green

SUMMARY:
The objective of this study is to determine if fluorescence lymphangiography can be used alone to localize sentinel nodes in patients with melanoma or breast cancer. The hypothesis is that sentinel nodes can be identified using only indocyanine green (ICG) and fluorescence lymphangiography, without the need for technetium99 and a gamma probe.

DETAILED DESCRIPTION:
From the subject's viewpoint, the course of events in this study will be no different than usual care and sentinel node biopsy. Subjects will have a dermal injection of technetium99 (tech99) at the melanoma tumor site prior to surgery (either the day before, or morning of surgery) or a subareolar injection if breast cancer. The surgeon will not look at the lymphoscintigraphy films, and the radiologist should not mark the skin. When the subject is in the operating room and appropriately sedated or anesthetized, tthey will receive a dermal injection of indocyanine green (ICG) 0.3-1.0 ml at the melanoma tumor site or subareola if breast cancer. Incision is made in the axilla or groin, and the SPY machine is positioned over the lymph node basin. Real-time lymphangiography (SPY) is used to identify sentinel nodes. Any fluorescent nodes should be resected and are considered sentinel nodes. The absolute fluorescence will be quantified for each sentinel node. Absolute fluorescence is calculated by the SPY machine.

After the sentinel lymphadenectomy is complete but prior to closing skin, the excised lymph nodes will be examined with the gamma probe (detects tech99 signal) to confirm that they are sentinel nodes. If the node does not have a signal with the gamma probe (but is fluorescent) it is still considered a sentinel node. The lymph node basin will also be examined with the gamma probe, to insure that no sentinel nodes are missed. If a gamma positive sentinel node is identified in the lymph node basin, it should be resected and imaged with SPY. If no sentinel nodes are able to be identified with fluorescent imaging, the gamma probe will be used as per usual practice. The surgeon should spend no more than 30 minutes using SPY to identify sentinel nodes. If after 30 minutes no sentinel node is found, the gamma probe should be used. The data collection form should be completed for each case.

The investigators intend to enroll at least 48 subjects. In order to insure that the data collected accurately represents the effectiveness of the SPY machine, each surgeon will be required to enroll at least 8 subjects into the study. Sentinel node biopsy is a routine surgical procedure, and all involved PIs are experienced in performing sentinel node biopsy. While fluorescence imaging intra-op is novel, the actual procedure itself is no different.

ELIGIBILITY:
Inclusion Criteria:

* Patients with melanoma or breast cancer who meet criteria for and consent to sentinel node biopsy.The melanoma should be located on the upper extremity between and including the wrist and shoulder, or the lower extremity between and including the ankle and groin.

Exclusion Criteria:

* Melanoma located on the trunk, head or neck. Patients with an allergy to indocyanine green or sodium iodide. Pregnant and nursing women. Patients who have had a prior sentinel node biopsy in the same nodal basin.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2017-10-11 (Actual); Primary Completion 2021-09-17 (Actual); Study Completion 2021-11-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Colette Pameijer, MD, Principal Investigator — Penn State Hershey Medical Center and College of Medicine
Locations (3):
- United States (3):
  - Emory University Hospital, Atlanta, Georgia
  - Vassar Brothers Medical Center, Poughkeepsie, New York
  - PennState Health Milton S. Hershey Medical Center, Hershey, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects recruited in surgical clinic between 10/11/2017 - 9/13/2021
Pre-assignment Details: One subject withdrew due to change in OR location and lack of SPY machine. No other relevant events.
Period: Overall Study
Arm/Group | Patients With Melanoma or Breast Cancer
Started | 35
Completed | 35
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Patients With Melanoma or Breast Cancer
Number analyzed (Participants) | 35
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 17
  >=65 years | 18
Age, Continuous [Mean (Full Range); unit: years] | 64.5 [28 to 88]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18
  Male | 17
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 0
  Unknown or Not Reported | 35
Region of Enrollment [Number; unit: participants]
  United States | 35
BMI [Mean (Full Range); unit: kg/m^2] | 27.3 [18.5 to 40.4]
Tumor location [Count of Participants; unit: Participants]
  Upper extremity | 21
  Lower extremity | 14

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Where the First, Second and Third Sentinel Nodes Localized With the Use of Fluorescence Imaging Alone
Description: The number of participants who had their first, second and third sentinel nodes correctly identified with ICG and fluorescence imaging alone, without the use of technetium99 and gamma probe. The number of sentinel nodes in any participant is determined by the patient's anatomy.
Time Frame: Intraoperative, up to 1 hour
Population: Patients with cutaneous melanoma of the extremity.
Measure: Count of Participants; unit: Participants
Arm/Group | Patients With Melanoma or Breast Cancer
Number analyzed (Participants) | 35
Participants
  First sentinel node | 29
  Second sentinel node: number analyzed (Participants) | 15
  Second sentinel node | 9
  Third sentinel node: number analyzed (Participants) | 5
  Third sentinel node | 0

2. Secondary Outcome: Adverse Events
Description: Any adverse events related to ICG or sentinel node biopsy.
Time Frame: Four weeks
Population: Patients with cutaneous melanoma of extremity who had a sentinel node biopsy
Measure: Number; unit: participants
Arm/Group | Patients With Melanoma or Breast Cancer
Number analyzed (Participants) | 35
participants | 7

ADVERSE EVENTS:
Time Frame: One month after surgery.
Description: Adverse events were collected intraop, postop and at the time of follow-up visit between 2-4 weeks after surgery.
Arm/Group | Patients With Melanoma or Breast Cancer
All-Cause Mortality (participants affected / at risk) | 0/35
Serious Adverse Events (participants affected / at risk) | 0/35
Other Adverse Events (participants affected / at risk) | 7/35
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Patients With Melanoma or Breast Cancer (N=35)
seroma (Skin and subcutaneous tissue disorders) | 3 (3)
hematoma (Skin and subcutaneous tissue disorders) | 2 (2)
SSI (Skin and subcutaneous tissue disorders) | 1 (1)
rash (Skin and subcutaneous tissue disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-05-27): https://cdn.clinicaltrials.gov/large-docs/30/NCT03294330/Prot_SAP_001.pdf